CLINICAL TRIAL: NCT03822676
Title: Prophylactic Pancreatic Stent for the Prevention of Post Operative Pancreatic Fistula Before Segmental Pancreatectomy
Brief Title: Prophylactic Pancreatic Stent for the Prevention of Post Operative Pancreatic Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZS-1833
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent (Experimental): Prophylactic pancreatic stent before segmental pancreatic surgery
  Interventions: Device: Prophylactic pancreatic stent
- No stent (No Intervention): No prophylactic stent before surgery

INTERVENTIONS:
Device: Prophylactic pancreatic stent — Prophylactic pancreatic stent before segmental pancreatic surgery
  Arms: Stent

SUMMARY:
Postoperative pancreatic fistula (POPF) remains one of the most harmful complications after pancreatic resection. Some studies have indicated that endoscopic pancreatic stenting was effective in the treatment of POPF. However, the results of prospective RCTs for the prophylactic effect of pancreatic stent insertion against POPF were controversial. This single center prospective randomized trial was designed to compare the outcome after segmental pancreatectomy with prophylactic drainage stent versus no stent.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective segmental pancreatectomy

Exclusion Criteria:

* Subjects for whom ERCP procedures are contraindicated
* If female, pregnant based on a positive hCG serum or an in vitro diagnostic test result or breast-feeding
* Age less than 18 year
* Emergency surgery
* Previous pancreatic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula | from postoperative day 3 to 30
  Grade B and C

SECONDARY OUTCOMES:
Severity of pancreatic fistula | from postoperative day 3 to 30
  Grade B POPF requires changes in clinical management, such as persistent drainage, partial or total parenteral nutrition, antibiotics, enteral nutrition, somatostatin analogs, and/or minimal invasive drainage. Grade C POPF requires major changes in management, such as admission to an intensive care unit, reoperation, and/or an extended hospital stay.
Length of stay | from postoperative day 1 to discharge
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China